CLINICAL TRIAL: NCT02811250
Title: Stereotactic Radiotherapy for Renal Cancers: Phase I Study
Brief Title: Stereotactic Radiotherapy for Renal Cancers
Acronym: RSR-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-556; 2010-A00087-32 (Other: ANSM)
Record Dates: First submitted 2016-06-08; First posted 2016-06-23 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Renal Cancer
Keywords: Renal cancer; Stereotactic radiotherapy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stereotactic radiotherapy 4 x 8 Gy (Experimental): Patient receive 4 stereotactic radiotherapy sessions with a dose of 8 Gy
  Interventions: Radiation: Stereotactic radiotherapy 4 x 8 Gy
- Stereotactic radiotherapy 5 x 8 Gy (Experimental): Patient receive 5 stereotactic radiotherapy sessions with a dose of 8 Gy
  Interventions: Radiation: Stereotactic radiotherapy 5 x 8 Gy
- Stereotactic radiotherapy 4 x 10 Gy (Experimental): Patient receive 4 stereotactic radiotherapy sessions with a dose of 10 Gy
  Interventions: Radiation: Stereotactic radiotherapy 4 x 10 Gy
- Stereotactic radiotherapy 4 x 12 Gy (Experimental): Patient receive 4 stereotactic radiotherapy sessions with a dose of 12 Gy
  Interventions: Radiation: Stereotactic radiotherapy 4 x 12 Gy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy 4 x 8 Gy
  Arms: Stereotactic radiotherapy 4 x 8 Gy
Radiation: Stereotactic radiotherapy 5 x 8 Gy
  Arms: Stereotactic radiotherapy 5 x 8 Gy
Radiation: Stereotactic radiotherapy 4 x 10 Gy
  Arms: Stereotactic radiotherapy 4 x 10 Gy
Radiation: Stereotactic radiotherapy 4 x 12 Gy
  Arms: Stereotactic radiotherapy 4 x 12 Gy

SUMMARY:
Stereotactic radiotherapy is a technique that allows the delivery of a high dose of radiation over few fractions (3-6) with great precision. It thus allows "tumor ablation" and optimal preservation of healthy tissues. Initially developed in small-sized (<5 cm) lung cancers this technique it gives results very close and or even equivalent to those of surgery.

Stereotactic radiotherapy of brain metastases of renal cancers has shown that high doses of radiation allows local control in 90 to 98% of cases. A study conducted in Sweden (Wersall et al.) underline the interest to develop stereotactic radiotherapy in primary renal tumors. In Cleveland (USA) two phase I studies are already underway.

The investigators propose to develop a phase I study for tumors of less than 4 cm. As found in lung cancers, stereotactic radiotherapy can provide a non-invasive, painless and rapid (4 to 5 fractions) method for the treatment of renal cancers with a high rate of local control.

The primary objective is to define the maximal tolerated dose for one fraction in stereotactic mode of renal tumors ≤ 4 cm in length using an a four-step dose increase:

* Step 1: 4 x 8 Gy.
* Step 2: 5 x 8 Gy.
* Step 3: 4 x 10 Gy.
* Step 4: 4 x 12 Gy.

The patients will be followed during treatment with evaluation of acute toxicities before each session, then at 15 days, 6 weeks, 3 months, 9 months, 12 months, and then every 6 months for a total duration of 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 75 years with an operable renal tumor or patient with inoperable renal tumor irrespective of age, or patient with metastatic renal tumor and indication for nephrectomy.
* Histologically-confirmed Renal carcinoma less than or equal to 4 cm
* Tumor that is visible and measureable on abdominal scanner and/or MRI (Magnetic Resonance Imaging)
* Karnofsky performance status ≥ 60%

Exclusion Criteria:

* Patient with only one kidney and renal cancer
* Patient not able to cooperate during treatment
* Previous history of abdominal radiation therapy
* Tumor having infiltrated the renal pelvis
* Polycystic kidney disease
* Previous history of intestinal inflammatory disease such as ulcerative colitis or Crohn's disease
* Renal insufficiency (creatinine clearance <30 ml/mm evaluated by DTPA (diethylenetriamine pentaacetic acid ) scintigraphy)
* Uncontrolled hypertension (SBP(systolic blood pressure) above 160 mmHg DBP(diastolic blood pressure) above 100 mmHg with antihypertensive treatment)
* Non primary lesions (benign lesions such as angiomyolipoma, renal metastases,…)
* Antineoplastic and/or antiangiogenic treatment in the month preceding radiotherapy
* Progressive cancer other than renal cancer at time of inclusion with the exception of in situ cervical carcinomas, basal cell carcinoma of the skin, and non-metastatic prostate cancer controlled without hormone therapy
* Participation in another ongoing study that may interfere with the present study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of grade ≥ 4 toxicity | 3 months after treatment
  The primary outcome is the occurrence of grade ≥ 4 toxicity according to CTCAE version 4 (Common Terminology Criteria for Adverse Events) during treatment and in the 3 months after end of treatment .

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Radiothérapie - Centre Georges François Leclerc, Dijon
  - Service d'Oncologie-Radiothérapie - Centre Hospitalier Lyon Sud - HCL, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lapierre A, Badet L, Rouviere O, Crehange G, Berthiller J, Paparel P, Chapet O. Safety and Efficacy of Stereotactic Ablative Radiation Therapy for Renal Cell Cancer: 24-Month Results of the RSR1 Phase 1 Dose Escalation Study. Pract Radiat Oncol. 2023 Jan-Feb;13(1):e73-e79. doi: 10.1016/j.prro.2022.06.012. Epub 2022 Jul 14. PMID 35842186